CLINICAL TRIAL: NCT01540981
Title: Multi-Center Study of the Effects of MIST Therapy on the Treatment of Deep Tissue Injury
Brief Title: Deep Tissue Injury Treatment With MIST Therapy Versus Standard Care: REVERSE DTI Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: Celleration, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CR-86034
Record Dates: First submitted 2012-02-20; First posted 2012-02-29 (Estimated); Results first posted 2014-12-15 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Wound of Skin
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SOC - Standard of Care (Active Comparator): Standard of care consists of pressure relief, creams, wound cleansing and dressings as needed
  Interventions: Other: Standard of Care
- MIST Therapy with SOC (Active Comparator): Standard of Care including pressure relief, wound cleansing, creams, and dressings as needed plus MIST Therapy daily for 5 days and then every other day for up to 7 more days
  Interventions: Device: MIST Therapy

INTERVENTIONS:
Device: MIST Therapy — FDA cleared non-contact ultrasound device. Delivers low frequency ultrasound via a fine saline to the wound area.
  Other Names: MIST Therapy, MIST, Non-Contact Ultrasound
  Arms: MIST Therapy with SOC
Other: Standard of Care — Standard of Care consists of pressure relief, wound cleansing and dressing as needed
  Arms: SOC - Standard of Care

SUMMARY:
The purpose of this study is to evaluate the effectiveness of MIST Therapy in conjunction with standard of care (SOC) compared to SOC alone in the prevention of deep tissue injury (DTI) progression to advanced stage pressure ulcers.

DETAILED DESCRIPTION:
Enrolled subjects will be randomized to receive one of two treatment courses: a) MIST Therapy in conjunction with Standard of Care (MIST + SOC) (treatment group) or b) SOC only (control group).

A randomized subject will be required to undergo a Baseline Evaluation. The Baseline Evaluation. A digital photo will be taken of the wound.

The subject will receive the assigned study treatment. Each subject will receive SOC wound care and off-loading daily throughout the study. Subjects will be treated daily for 5 days and then every other day until discharged or up to 14 days post enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject of any race 18-90 years old.
* Subject presents with an index DTI. This is defined by the National Pressure Ulcer Advisory Panel (NPUAP) as a purple or maroon localized area of discolored intact skin or blood-filled blister due to damage of underlying soft tissue from pressure and/or shear. The area may be preceded by tissue that is painful, firm, mushy, boggy, warmer or cooler as compared to adjacent tissue.
* Subject's DTI has been discovered ≤ 72 hours after causative event
* Causative event of DTI is identified.
* Subject's index DTI is located on torso or body extremities.
* Subject is currently admitted to the hospital.
* Subject is able to be maneuvered into a position that is acceptable for MIST treatment.
* Subject's DTI presents with no clinical signs of acute infection.
* Subject or subject's legally authorized representative understands the nature of the procedures and provides written informed consent prior to study enrollment.

Exclusion Criteria:

* Subject's primary wound is a Stage I, Stage II, Stage III or Stage IV pressure ulcer.
* Subject's wound presents with a malignancy in the wound bed.
* Subject has a history of pressure ulcer / DTI in same location.
* Subject's DTI would require ultrasound near an electronic implant or prosthesis, e.g., near or over the heart, or over the thoracic area if the patient is using a cardiac pacemaker.
* Female subjects that are pregnant or refuse to utilize adequate contraceptive methods and are of childbearing age during the trial.
* Subject is terminally ill, defined as unable to survive beyond 14 days.
* Subject is known to be suffering from a disorder or other situation that the subject or investigator feels would interfere with compliance or other study requirements.
* Subject is currently enrolled or has been enrolled in the last 30 days in another device or drug trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2013-06 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Black, PhD, RN, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SOC - Standard of Care | MIST Therapy With SOC
Started | 6 | 6
Completed | 5 | 6
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SOC - Standard of Care | MIST Therapy With SOC | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Median (Full Range); unit: years] | 55 [28 to 77] | 69.5 [62 to 77] | 65 [28 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11
BMI [Median (Full Range); unit: kilograms per meter squared] — kilograms per meter squared
  kilograms per meter squared | 28.6 [22.2 to 55.4] | 27.7 [24.4 to 45.4] | 28.6 [22.2 to 55.4]
Type of Injury Leading to Suspected DTI [Number; unit: participants]
  Sustained Immobility | 1 | 5 | 6
  Shearing | 1 | 0 | 1
  Cardiac Arrest/Hemodynamic Crash | 1 | 0 | 1
  Other | 2 | 1 | 3
Wound Size [Median (Full Range); unit: centimeters squared] — Wound area measured as centimeters squared
  centimeters squared | 3.8 [0.6 to 10.0] | 13.9 [1.0 to 168.8] | 7.4 [0.6 to 168.8]
Wound Location [Number; unit: participants]
  Heel | 1 | 2 | 3
  Ischium | 0 | 1 | 1
  Sacrum/Coccyx | 4 | 2 | 6
  Buttocks | 0 | 1 | 1
Age of Wound [Median (Full Range); unit: days] | 3.0 [1.0 to 5.0] | 2.5 [0 to 4] | 3.0 [0 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness
Description: To compare between the treatment groups the effect of the assigned study treatment on the rate of progression of DTI to advanced stage pressure ulcer (Stage III or greater, continued DTI, or a pressure ulcer that is unable to be staged due to necrotic tissue).
  Stage I - Intact skin with non-blanchable redness of a localized area Stage II - Partial thickness loss of dermis Stage III - Full thickness loss, subcutaneous fat may be visible Stage IV - Full thickness tissue loss with exposed bone, tendon or muscle Unstageable - Full thickness tissue loss in which the base of the ulcer is covered by slough or eschar Continues deep tissue injury - purple or maroon localize area of discolored intact skin that may be mushy or boggy
Time Frame: 14 days
Measure: Number; unit: participants
Arm/Group | SOC - Standard of Care | MIST Therapy With SOC
Number analyzed (Participants) | 5 | 6
participants
  Healed | 0 | 1
  Pressure Ulcer Stage II | 1 | 1
  Unstageable | 0 | 2
  DTI | 4 | 2

2. Secondary Outcome: Change in Mean Wound Area
Description: Measured from randomization to last visit (14 days or at discharge from hospital)
Time Frame: 14 days
Measure: Mean (Standard Deviation); unit: square centimeters
Arm/Group | SOC - Standard of Care | MIST Therapy With SOC
Number analyzed (Participants) | 5 | 6
square centimeters | 0.94 (6.54) | -21.5 (42.4)

ADVERSE EVENTS:
Time Frame: Study duration 14 days
Arm/Group | SOC - Standard of Care | MIST Therapy With SOC
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6

LIMITATIONS AND CAVEATS:
Follow-up limited by discharge from hospital.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No